CLINICAL TRIAL: NCT04328935
Title: A Feasibility Study for Written Exposure Therapy for Patients With Post-traumatic Stress Disorder in a Regular Health Care Setting
Brief Title: Written Exposure Therapy for Post-traumatic Stress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Erik Andersson, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-04414
Record Dates: First submitted 2020-03-15; First posted 2020-04-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; written exposure therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Within-group design. Repeated measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- written exposure therapy (Experimental): The treatment consists of written exposure therapy (WET), which is manualized trauma-focused CBT in five sessions over 5 weeks.
  Interventions: Behavioral: WET

INTERVENTIONS:
Behavioral: WET — The manual is based on established CBT interventions in trauma such as exposure. In short, the treatment is that the participant should be able to approach their intrusive memories and by doing this repeatedly, the memory will give rise to less discomfort.

SUMMARY:
To investigate if written exposure therapy is feasible for patients with post-traumatic stress disorder

DETAILED DESCRIPTION:
A non-inferiority trial in JAMA Psychiatry showed that written exposure therapy (WET) was non-inferior to a gold standard CBT treatment. In comparison to other trauma-focused CBT protocols, WET generally demands less therapist-time, and specifically, less than half compared to CBT that consists of 12 weekly sessions á 60 minutes. The aim of this study is to translate and replicate these results in a Swedish context. This first step is a small feasibility trial which will guide a subsequent large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for PTSD.
* If taking psychotropic medication, then the dose must be stable for at least 4 weeks prior to study entry.
* ≥ 18 years
* Situated in Sweden
* Be able to express themselves in Swedish, both in verbally and written form.
* Informed consent

Exclusion Criteria:

* Other serious comorbidity as primary concern (ongoing substance dependence, untreated bipolar disorder, psychotic symptoms, severe depression, borderline personality disorder, high suicidal risk according to the MINI)
* Ongoing CBT for trauma
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-04-27 (Estimated)

PRIMARY OUTCOMES:
The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Time Frame: Baseline, week 5 and follow-up at 6 months
  Change in symptoms of post traumatic stress from baseline to post treatment and follow up (6 months). The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms. All items are scored on a 0-4 scale. Higher score indicate worse severity

SECONDARY OUTCOMES:
Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) | Time Frame: Baseline, week 5 and follow-up at 6 months
  Change in depressive symptoms from baseline to post treatment and follow up (6 months). The Montgomery Åsberg Depression Rating Scale - Self-report (MADRS-S) is a 9 item self-report measure that assesses the presence and severity of depressive symptoms. All items are scored on a 0-6 scale. Higher score indicate worse severity.
Euroqol, EQ-5D | Time Frame: Baseline, week 5 and follow-up at 6 months
  Change in overall health from baseline to post treatment and follow up (6 months). EQ-5D is a standardised self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Case report form (CRF) data will be imputed to a data file. Analysis will be performed by members of the study-team and quality control and crosscheck will be performed by independent party.

REFERENCES:
- [Derived] Hedvall H, Andersson E, Ivanov VZ, Bragesjo M. Feasibility of written exposure therapy for PTSD in a psychiatric outpatient clinic: in-person and remote delivery. Eur J Psychotraumatol. 2025 Dec;16(1):2545048. doi: 10.1080/20008066.2025.2545048. Epub 2025 Sep 2. PMID 40891431